CLINICAL TRIAL: NCT01661517
Title: Brief Intervention and Referral to Treatment With Substance Use Disorders in the Emergency Room Setting (Screening and Brief Treatment for Substance Use Disorders in the Emergency Room Department)
Brief Title: Brief Intervention and Referral to Treatment With Substance Use Disorders in the Emergency Room Setting
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: incomplete data
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: X110829003
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-09

CONDITIONS: Substance Use
Keywords: substance use treatment
MeSH Terms: conditions — Substance-Related Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle Counseling (Experimental): motivational interviewer
  Interventions: Behavioral: Motivational interviewing and referral to treatment

INTERVENTIONS:
Behavioral: Motivational interviewing and referral to treatment

SUMMARY:
This study will be a quality improvement project to review the effectiveness and barriers to effectiveness of a new clinical program in the emergency room to provide substance use screening followed by brief motivational interviewing and referral to treatment for patients who meet criteria for problem substance use. This study will consist of a chart review of the results of the screens performed by substance use counselors and correlating them to institutional variables such as wait time in the emergency room and length of stay as well as to patient variables obtained by chart review such as medical diagnosis and sociodemographic variables.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 and older Presentation to UAB Emergency Department

Exclusion Criteria:

* Younger than 19 Prisoners

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5271 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
substance use | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama Birmingham, Birmingham, Alabama, United States